CLINICAL TRIAL: NCT04749017
Title: A Double Blind, Randomized, Controlled Study for the Potential Effect of Avena Sativa L. on Wellness/Wellbeing During Smoking Reduction/Cessation Experience
Brief Title: The Potential Effect of Avena Sativa L. on Wellness/Wellbeing During Smoking Reduction/Cessation Experience
Acronym: SMOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00018
Record Dates: First submitted 2020-12-01; First posted 2021-02-10 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-10

CONDITIONS: Smoking Reduction
Keywords: Wellbeing; Wellness
MeSH Terms: conditions — Smoking Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Avena Sativa L. consumption of 900 mg for 60 days.
  Interventions: Dietary Supplement: Experimental product consumption
- Control group (Placebo Comparator): Identically appearing placebo capsules consumed for 60 days.
  Interventions: Other: Control product consumption

INTERVENTIONS:
Dietary Supplement: Experimental product consumption — Consumption of the experimental product 2 capsules daily, morning and evening (450 mg each capsule) for 60 days
  Arms: Experimental group
Other: Control product consumption — Consumption of control product of identical appearance 2 capsules daily for 60 days, morning and evening
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the potential effect of Avena Sativa L. on wellbeing during smoking reduction/cessation

DETAILED DESCRIPTION:
The duration of the study will be 90 days (12 weeks). The consumption time will be set at 60 days (8 weeks), the remaining 30 days will be for follow up, the product will not be consumed. Each day of the study will be recorded in a diary by each subject.

Subjects are randomized based on the number of cigarettes and the Richmond test. In addition, subjects with a high score on the DASS-21 test items could not participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age: 18 - 65 YO)
* Willingness to reduce/quit daily cigarettes (Richmond test)
* Regular smokers: ≥10 CPD for the last 6 months (mean of ~16)
* At least 6 months of smoking
* Exhaled CO level≥10 ppm
* Healthy adults:

  1. Normal blood profile at screening
  2. Subject is in a good physical health as established by medical history, vital signs, self-declaration and physical examination
  3. Without depression/ anxiety or stress (based on a psychological evaluation and DASS21 questionnaire)
* Able to participate fully in all aspects of the study and had understood and signed the informed consent
* Negative drug test (THC, Amphetamines, Methamphetamines, Cocaine and Opioids)
* For women: Negative pregnancy test

Exclusion Criteria:

* Use of any mineral/vitamin/drug or other supplements during the past month prior to study
* Participate in another clinical trial in the last 6 months
* Using (past 30 days) other smoking cessation aids, for example treatments for tobacco dependence or an investigational drug
* Smoke other nicotine-containing products such as hookah smokeless tobacco or electronic cigarettes
* Allergic or intolerance to one of the ingredients of the investigated product
* Diagnosed or treated for mental illness/ disorder in the past year
* Recent history (past year) of alcohol or drug abuse or dependence
* Reported any active/chronic disease (such as: Celiac disease/active peptic ulcer) or chronic medications (except Hyperlipidaemia or hypertension that are stable on medications)
* Any other laboratory abnormality, medical condition or psychiatric disorder which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
* Pregnant, lactating women or women that plan to get pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Wellbeing / wellness | From baseline to 8 weeks later
  WHOQOL BREF test

SECONDARY OUTCOMES:
Wellbeing / wellness | Day 1, at 4 and 12 weeks later
  WHOQOL BREF test
Cognitive performance | Day 1, at 4, 8 and 12 weeks later
  COMPASS cognitive test panel
Quality of life panel | Day 1, at 4, 8 and 12 weeks later. They also have to fill it in at home, in a diary, on the 15th, 45th and 75th day.
  Using a visual analog scale where 0=not good at all, 10=very good
Quality of life questionnaire | Day 1, at 4 and 8 weeks later
  SF-36 test health questionnaire
Brief questionnaire of smoking urges | Day 1, at 4 and 8 weeks later
  QSU-Brief/Tiffany test
Depression | Day 1, at 4 and 8 weeks later
  Beck depression. Test to measure the level of depression of the subjects
Perceived stress scale | Day 1, at 4 and 8 weeks later
  Scale Remor, 2001. Test to measure the level of stress of the subjects
Anxiety questionnaire | Day 1, at 4 and 8 weeks later
  Test STAI, to measure the level of anxiety of the subjects
Biopyrrin | Day 1, at 4 and 8 weeks later
  Measured in urine
Cortisol | Day 1, at 4 and 8 weeks later
  Measured in saliva
Nicotine Dependence | Day 1, at 4 and 8 weeks later
  Fagerstrom test (FTND)
Minnesota Nicotine Withdrawal scale | Day 1, at 4 and 8 weeks later
  Nicotine withdrawal scale
Number of cigarettes per day | Number of daily cigarettes is recorded on a daily basis in the diary from week 1 to week 12. Cotinine and exhaled carbon moxide are measured on day 1, at 4, 8 and 12 weeks later
  Cigarettes per day self-reported in the daily diary, validated by cotinine and exhaled carbon monoxide at every visit
Craving level quantification | Day 1, at 4 and 8 weeks later
  Visual analog scale where 0=no desire to smoke, 10=strong desire to smoke
VAS symptoms severity panel | Day 1, at 4, 8 and 12 weeks later.
  Using a visual analog scale where 0=very low, 10=very high
Sleep efficiency | It will be measured during 3 weekdays and one weekend day, before starting with the consumption of the product and before the end of the consumption (60 days).
  Measured by accelerometry, with Actigraph wGT3X-BT

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

REFERENCES:
- [Derived] Friling M, Garcia-Munoz AM, Lavie A, Perez-Pinero S, Victoria-Montesinos D, Lopez-Roman FJ, Garcia-Guillen AI, Munoz-Carrillo JC, Canovas F, Ivanir E, Jalanka J. Dietary supplementation with a wild green oat extract (Avena sativa L.) to improve wellness and wellbeing during smoking reduction or cessation: a randomized double-blind controlled study. Front Nutr. 2024 Jun 19;11:1405156. doi: 10.3389/fnut.2024.1405156. eCollection 2024. PMID 38962436